CLINICAL TRIAL: NCT05999669
Title: Assessing the Predictive Value of the Global Limb Anatomic Staging System (GLASS) in EndoVascular Therapy (EVT) of Infrainguinal Lesions in Patients With Critical Limb-threatening Ischemia (CLTI): the GLASS-EVT Study
Brief Title: Predictive Value of the Global Limb Anatomic Staging System (GLASS) in Patients With Critical Limb-threatening Ischemia
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Second Affiliated Hospital of Soochow University (Other); First Affiliated Hospital of Zhejiang University (Other); First People's Hospital of Hangzhou (Other); Qingdao Haici Hospital (Other); Liyuan Hospital of Tongji Medical College, Huazhong University of Science and Technology (Other); Fudan University (Other); Huashan Hospital (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: GLASS-EVT
Record Dates: First submitted 2023-07-30; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Peripheral Arterial Disease
Keywords: global limb anatomic staging system; infrainguinal Lesion; critical limb-threatening ischemia
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: GLASS staging — use the Global Limb Anatomic Staging System (GLASS) to evaluate its correlation with clinical outcomes after revascularization

SUMMARY:
The Global Vascular Guideline on chronic limb threatening ischemia (CLTI) proposes the Global Limb Anatomic Staging System (GLASS), a new angiographic scoring system to quantify the anatomic severity of infrainguinal disease in CLTI patients. However, GLASS validation still needs to be completed, and the infrapopliteal (IP) target artery pathway (TAP) was easily influenced by the procedures. Thus the IP target artery could be selected either as the least diseased artery based on angiography or prospectively based on the angiosome concept. So the investigators aim to evaluate its correlation with clinical outcomes after revascularization.

DETAILED DESCRIPTION:
The Global Vascular Guideline on chronic limb threatening ischemia (CLTI) recommends using the Global Limb Anatomic Staging System (GLASS) to assess the severity of infrainguinal disease in CLTI patients. GLASS staging involves scoring the femoropopliteal (FP) and infrapopliteal (IP) segments separately. For IP segment scoring, the target artery path (TAP) is identified by the clinician based on either the least diseased or the recanalized IP path. However, this approach may lead to diverse GLASS staging results, especially for simple lesions below the knee. Additionally, the current version of GLASS does not account for multivessel IP revascularization, which may introduce subjective bias if a physician chooses different IP targets during multiple revascularization procedures.

In order to improve our understanding of the current staging system, the investigators will establish a prospective registry that collects data on conservative patients who have Chronic Limb-Threatening Ischemia (CLTI) and undergo endovascular therapy for infrainguinal lesions. To evaluate the stage of the lesions, the investigators will use two distinct IP scoring techniques. One approach will be based on the least disease IP path as identified by the pre-interventional angiogram, while the second technique will be based on the recanalized IP path preferred by the clinician. This scoring will be carried out by experienced physicians and the results will be recorded in an electronic database. Then the correlation between the major adverse limb events (such as clinical-driven target limb revascularization, major amputation, and all-cause death) with the patient's Wound, Ischemia, foot Infection (WIFI) classification, GLASS anatomic staging, calcification severity, and modified Society for Vascular Surgery (SVS) run-off score will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of chronic limb-threatening ischemia (CLTI)
2. Undergo endovascular therapy for infrainguinal lesions

Exclusion Criteria:

1. Pregnant women or female patients with potential childbearing
2. Patients who have acute limb thromboembolism or require thrombectomy during the procedure
3. Untreated inflow disease of the ipsilateral pelvic arteries (more than 50% stenosis or occlusion)
4. Patients with known allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with infrainguinal lesions suffering from critical limb-threatening ischemia
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-08-20 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of freedom from major adverse events (MAEs) | 12-month
  Major adverse events (MAEs) is defined as index limb amputation above the ankle, clinical-driven target lesion revascularization (CD-TLR), or all-cause death

SECONDARY OUTCOMES:
Rate of acute procedure success | 72-hour after procedure
  Acute procedure success is defined as technique success ( the achievement of final residual diameter stenosis <30% for stent and <50% for angioplasty or atherectomy by angiography at the end of the procedure and without flow-limiting arterial dissection or hemodynamically significant trans-lesional pressure gradient <10 mm Hg for endovascular revascularization ) and freedom form MAEs within 72 hours of the index procedure.
Rate of freedom from clinical-driven target lesion revascularization (CD-TLR) | 24-month
  Patients without clinical-driven target lesion revascularization (CD-TLR)
Rate of freedom from major adverse events (MAEs) | 24-month
  Major adverse events (MAEs) is defined as index limb amputation above the ankle, clinical-driven target lesion revascularization (CD-TLR), or all-cause death
Primary sustained clinical improvement assessed by Rutherford classification | 24-month
  Primary sustained clinical improvement is defined as an upward shift on the Rutherford classification to a level of claudication without the need for repeated target lesion revascularization in surviving patients without the need for unplanned amputation.
Change of quality of life assessed by Vasc quality of life scale | 24-month
  Postoperative Vasc quality of life score minus preoperative Vasc quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ye, M.D., Principal Investigator — Department of Vascular Surgery, Renji Hospital, School of Medicine, Shanghai Jiaotong University

IPD SHARING:
Plan to Share IPD: Undecided